CLINICAL TRIAL: NCT06102291
Title: Effect of Acupoint Application With Yanqing Zhitong Ointment for Chronic Non-specific Low Back Pain: a Non-inferiority Randomized Controlled Trial
Brief Title: Acupoint Application With Yanqing Zhitong Ointment for Chronic Non-specific Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZhanYJ (Other)
Responsible Party: Sponsor-Investigator, ZhanYJ, Shanghai University of Traditional Chinese Medicine, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YD202218
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Non-specific Low Back Pain
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupoint application with Yanqing Zhitong Ointment (Experimental): Acupoint selection: Ashi points, Shenshu (BL23), Guanyuanshu (BL26) Operation: Stick to each acupoint for about 4 hours. If there is a burning sensation or obvious itching or other discomfort on the part after application, it can be removed in advance.
  Treatment Duration: Three times a week( Monday, Wednesday, and Friday), for four weeks
  Interventions: Other: Yanqing Zhitong Ointment Acupoint application
- Acupuncture (Active Comparator): Acupoint selection: Ashi points, Shenshu (BL23), Guanyuanshu (BL26) Operation: Disposable stainless steel needles (0.25mm×25mm) are used. The needles are retained for 20 mins afte Deqi.
  Treatment Duration: Three times a week( Monday, Wednesday, and Friday), for four weeks
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Yanqing Zhitong Ointment Acupoint application — Yanqing Zhitong Ointment is a traditional external preparation of experiential prescription, which is an extract made by water extraction and concentration of Qingfengteng, Corydalis yanhusuo, Interleukin, Kansui, Asarum, etc. Clinical studies in the past ten years have preliminarily shown that it has the effects of warming meridians, promoting blood circulation, dredging collaterals and relieving pain, and has a definite effect.
  Arms: Acupoint application with Yanqing Zhitong Ointment
Other: Acupuncture — The main acupoints are Ashi points, Shenshu (BL23), Guanyuanshu (BL26). There are three sessions per week with each session lasting for 20 min. There will be 4 weeks of treatment for each participant in total.
  Arms: Acupuncture

SUMMARY:
This is a non-inferiority randomized controlled trial, recruiting 150 patients with chronic non-specific low back pain. The patients will be randomly assigned either to Yanqing Zhitong Ointment acupoint application group (Treatment Group) or the acupuncture group (Control Group) in a 1:1 ratio.

DETAILED DESCRIPTION:
This is a non-inferiority randomized controlled trial, 150 patients with chronic non-specific low back pain were randomly assigned to acupoint application group and acupuncture group in a 1:1 ratio. The main acupoints are Ashi points, Shenshu(BL23), Guanyuanshu(BL26). The primary outcome measure is the change of McGill Pain Questionnaire (MPQ) before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with non-specific low back pain
2. Aage from 18 to 65
3. VAS between 4 and 7
4. No other treatment in the past 3 months
5. No other simultaneous relevant treatment
6. Voluntarily joining this study with informed consents

Exclusion Criteria:

1. Pregnant women
2. With skin ulcers or contusion wounds
3. Past history of severe allergy to transdermal preparations
4. Complicated with serious diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
McGill pain questionnaire | Change from baseline to Week 4
  MPQ is a multi-factor pain score scale, which establishes a three-dimensional structure of the nature of pain. MPQ has a higher evaluation dimension and can evaluate the multi-dimensional factors of pain. The higher the score, the more severe the pain.

SECONDARY OUTCOMES:
McGill pain questionnaire | Change from baseline to Week 8 (follow-up)
  MPQ is a multi-factor pain score scale, which establishes a three-dimensional structure of the nature of pain. MPQ has a higher evaluation dimension and can evaluate the multi-dimensional factors of pain. The higher the score, the more severe the pain.
Oswestry Dysfunction Index (ODI) | Change from baseline to Week 4 and Week 8
  ODI is a self-evaluation scale for dysfunction of patients with low back pain. It consists of 10 aspects including pain degree, personal living ability (washing, dressing), lifting, walking, sitting, standing, sleep influence, sex life, social activities and travel. Each aspect covers 6 options, with points ranging from 0 to 5 points. The lowest score indicates no abnormal dysfunction, and the highest score indicates severe dysfunction. The corresponding candidate content scores are added up in turn according to the scores, and the percentage of the total score in the highest score (50 points) of all content is obtained, which is called the Oswe-stry dysfunction index.
Item Short Form Health Survey (SF-36) | Change from baseline to Week 4 and Week 8
  SF-36 is currently one of the most widely used universal health-related quality of life measurement tools in the world. SF-36 covers 8 dimensions for assessing health-related quality of life and a total of 36 content items. Each dimension includes: physical function (PF), role physical (RP), bodily pain (BP), General health (GH), vitality (VT), social function (SF), role-emotional (RE) and mental health (MH). SF-36 first calculates the original scores of the eight dimensions, and then obtains the final score after corresponding conversion. The final score is 0-100 points. The higher the final score, the better the health of the testee.
Tenderness threshold | Change from baseline to Week 4 and Week 8
  Use the digital pressure pain meter to measure the pressure pain threshold of soft tissues and muscles, and conduct an objective and quantitative assessment of pain. It is used for auxiliary diagnosis and scientific research of pain in muscles and tendons.

CONTACTS AND LOCATIONS:
Overall Officials: Yijun Zhan, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, China

REFERENCES:
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Wen BL, Liu BY, Jin P, Wang XF, Xiang XX, Liu XF, Hu JQ, Lu F, He LY, Zhu WZ, Fang YG, Wang Y. Clinical research of acupoint application for "treatment of winter disease in summer" used to prevent and treat bronchial asthma in children. J Tradit Chin Med. 2012 Mar;32(1):31-9. PMID 22594099